CLINICAL TRIAL: NCT01797757
Title: Comparison of the Efficacy of Monoacylglycerol (MAG) and Triacylglycerol (TAG) to Deliver Long Chain Polyunsaturated Fatty Acids (LC-PUFA) Under Malabsorption Conditions
Brief Title: Comparison of MAG and Fish Oil Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 10.29.NRC
Record Dates: First submitted 2013-02-19; First posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Obesity
Keywords: EPA; LC-PUFA; Orlistat; Obesity
MeSH Terms: conditions — Obesity | interventions — 1-eicosapentaenoylglycerol; Orlistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fish oil enriched with EPA + ORLISTAT (Active Comparator): The oil will be liquid form of 1g /capsule. 3 capsules will be administrated per day: one capsule to be swallowed with a glass of water before every major meal, 3 times a day for 21 days.
  The Orlistat capsules of 120mg (except for groups 1 and 2). 3 capsules will be administrated per day: one capsule to be swallowed with a glass of water before every major meal, 3 times a day for 21 days.
  Interventions: Dietary Supplement: Fish oil enriched with EPA; Drug: Orlistat
- MAG-EPA (Active Comparator): The oil will be liquid form of 1g /capsule. 3 capsules will be administrated per day: one capsule to be swallowed with a glass of water before every major meal, 3 times a day for 21 days.
  Interventions: Dietary Supplement: MAG-EPA oil
- MAG-EPA + ORLISTAT (Active Comparator): The oil will be liquid form of 1g /capsule. 3 capsules will be administrated per day: one capsule to be swallowed with a glass of water before every major meal, 3 times a day for 21 days.
  The Orlistat capsules of 120mg (except for groups 1 and 2). 3 capsules will be administrated per day: one capsule to be swallowed with a glass of water before every major meal, 3 times a day for 21 days.
  Interventions: Dietary Supplement: MAG-EPA oil; Drug: Orlistat
- Fish oil enriched with EPA (Active Comparator): The oil will be liquid form of 1g /capsule. 3 capsules will be administrated per day: one capsule to be swallowed with a glass of water before every major meal, 3 times a day for 21 days.
  Interventions: Dietary Supplement: Fish oil enriched with EPA

INTERVENTIONS:
Dietary Supplement: Fish oil enriched with EPA
  Arms: Fish oil enriched with EPA; Fish oil enriched with EPA + ORLISTAT
Dietary Supplement: MAG-EPA oil
  Arms: MAG-EPA; MAG-EPA + ORLISTAT
Drug: Orlistat
  Arms: Fish oil enriched with EPA + ORLISTAT; MAG-EPA + ORLISTAT

SUMMARY:
A potential application for unstructured monoacylglycerol (MAG) containing long chain polyunsaturated fatty acids (LC-PUFA)can be to provide essential fatty acids to humans who chronically consume lipases inhibitor such as Orlistat® for weigh lowering reasons. Indeed, it is predictable that chronic consumption of Orlistat® led to a depletion of essential fatty acids with time, therefore unstructured MAG containing LC-PUFA can be an option as a source of LC-PUFA for patients under Orlistat® treatment and hypothetically for subjects with other type of maldigestion/malabsorption. Potential applications of such concept are therefore related to disease conditions comprising low lipid digestion due to lipase activity insufficiency.

In the present study, in order to see the response information for eicosapentanoic acid (EPA) delivery, EPA will be provided either as a mixture of free monoacylglycerols or as triacylglycerol (TAG). The erythrocyte and plasma fatty acid composition from subjects under Orlistat® consumption will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Sex female
* Body Mass Index (BMI) ≥ 30kg/m2 and < 40kg/m2
* Subjects willing to undergo treatment with Orlistat® (Xenical).
* Having obtained her written informed consent before any study related procedure including the pre-inclusion period.

Subject exclusion criteria:

* Binge eating disorder
* Any other weight loss treatment(s) within the last 3 months
* Vegetarians
* History of metabolic, cardiovascular, hepatic or renal diseases
* Obstructed bile duct
* Diseases that could interfere with intestinal absorption History of abdominal / gastric surgery (except appendicectomy)
* Use of drugs or illicit substances
* Consumption of alcohol > 50 gr/week
* Any other clinically significant abnormalities on screening laboratory evaluation (creatinine, Na, K, urique acide, ASAT, ALAT, Ph. Alc., yGT, Glycemia, total cholesterol, HDL, LDL, triglycerides) concentrations > 2.5 fold normal range
* Pregnant or lactating mothers
* Allergy to fish oil or other components (for e.g., gelatin or excepients of the capsule)
* Use of any other supplements containing fish oil for the duration of the trial or 3 month before inclusion in trial.
* Smokers
* Having donated blood or had a transfusion of blood/blood products during the trial and 3 months prior to screening or expected to do so during the study
* Bleeding disorders
* Subject who cannot be expected to comply with the study procedures.
* Currently participating or having participated in another clinical trial during last 8 weeks prior to the beginning of this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be accretion of EPA in erythrocytes at 21days | 21 days

SECONDARY OUTCOMES:
• The secondary outcome will be the incorporation of EPA in plasma + chylomicrons | from baseline to day 21

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Giusti, MD, Principal Investigator — CHUV Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUV Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Cruz-Hernandez C, Destaillats F, Thakkar SK, Goulet L, Wynn E, Grathwohl D, Roessle C, de Giorgi S, Tappy L, Giuffrida F, Giusti V. Monoacylglycerol-enriched oil increases EPA/DHA delivery to circulatory system in humans with induced lipid malabsorption conditions. J Lipid Res. 2016 Dec;57(12):2208-2216. doi: 10.1194/jlr.P070144. Epub 2016 Oct 5. PMID 27707818